CLINICAL TRIAL: NCT01514149
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Phase 2 Dose-Ranging Study to Evaluate the Efficacy and Safety of 17 Weeks of Weekly Injections of CJC-1134-PC in Patients With Type 2 Diabetes Mellitus on Metformin Monotherapy
Brief Title: Dose-Ranging Study to Evaluate Efficacy and Safety of Weekly CJC-1134-PC in Patients With T2DM on Metformin Monotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: ConjuChem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DM200-103
Record Dates: First submitted 2011-10-20; First posted 2012-01-20 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Type 2 Diabetes Mellitus; T2DM; diabetes; ConjuChem; GLP-1; Glucagon-like peptide-1; exendin-4; modified exendin-4
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 - Weekly CJC-1134-PC (Experimental)
  Interventions: Drug: CJC-1134-PC Injection
- Arm 2 - Weekly CJC-1134-PC (Experimental)
  Interventions: Drug: CJC-1134-PC Injection
- Arm 3 - Weekly CJC-1134-PC (Experimental)
  Interventions: Drug: CJC-1134-PC Injection
- Arm 4 - Weekly CJC-1134-PC (Experimental)
  Interventions: Drug: CJC-1134-PC Injection
- Arm 5 - Weekly Placebo (Placebo Comparator)
  Interventions: Drug: Weekly placebo for CJC-1134-PC Injection

INTERVENTIONS:
Drug: CJC-1134-PC Injection — CJC-1134-PC administered weekly by subcutaneous injection
  Other Names: metformin
  Arms: Arm 1 - Weekly CJC-1134-PC; Arm 2 - Weekly CJC-1134-PC; Arm 3 - Weekly CJC-1134-PC; Arm 4 - Weekly CJC-1134-PC
Drug: Weekly placebo for CJC-1134-PC Injection — Weekly placebo for CJC-1134-PC administered weekly by subcutaneous injection
  Other Names: metformin
  Arms: Arm 5 - Weekly Placebo

SUMMARY:
DM200-103 is a dose-ranging study to evaluate the efficacy and safety of 17 weeks of weekly injections of CJC-1134-PC in patients with Type 2 Diabetes Mellitus on metformin monotherapy.

DETAILED DESCRIPTION:
DM200-103 is a dose-ranging study to evaluate the efficacy and safety of 17 weeks of weekly injections of CJC-1134-PC in patients with Type 2 Diabetes Mellitus (T2DM) on metformin monotherapy. This study will be a randomized, double-blind comparison of CJC-1134-PC versus placebo. Patients taking metformin will continue to take their metformin at the same dose for the duration of the study.

Patients with T2DM, who meet all the inclusion criteria and none of the exclusion criteria, will be randomly assigned to a treatment arm. All patients will undergo weekly clinic visits to receive 17 weeks of study treatment, including the titration period.

CJC-1134-PC or placebo treatment will be administered weekly by subcutaneous injection in the abdomen to patients in a fasting state. Patients will be closely monitored and evaluated for toxicity on an ongoing basis.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 to 70 years of age, inclusive
* Body mass index of 27 to 45 kg/m2
* Diagnosed with T2DM for at least 6 months before screening
* Stable daily dose of metformin monotherapy of ≥1000 mg for at least 3 months before screening
* FPG ≤240 mg/dL at screening
* HbA1c ≥7.0% and ≤11% at screening
* A 12-lead electrocardiogram recording without clinically significant arrhythmia, left bundle-branch block, or corrected QT interval

Exclusion Criteria:

* Pregnant or breastfeeding women
* Use of a weight control treatment, including over-the-counter medications (includes herbal supplements), or a significant change in body weight (at least ±10%) in the 3 months before screening
* Treatment with any oral antidiabetic agent other than metformin within the 3 months before screening
* Treatment with insulin for longer than 1 week within the 3 months before screening or any treatment with insulin within the 2 weeks before screening
* Previous treatment with a glucagon-like peptide 1 (GLP-1) analog or other incretin therapy
* Receipt of any experimental drug in a clinical trial within 30 days before administration of study drug or receipt of any investigational antidiabetic product within 3 months before screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Soon-Shiong, MD, Study Director — Chief Executive Officer; Robert Henry, MD, Principal Investigator
Locations (22):
- United States (19):
  - Research Site, Phoenix, Arizona
  - Research Site, Inglewood, California
  - Research Site, Tarzana, California
  - Research Site, Ventura, California
  - Research Site, Wellington, Florida
  - Research Site, Idaho Falls, Idaho
  - Research Site, Lexington, Kentucky
  - Research Site, Brighton, Massachusetts
  - Research Site, Greensboro, North Carolina
  - Research Site, Eugene, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Taylors, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Henrico, Virginia
- Canada (3):
  - Research Site, Vancouver, British Columbia
  - Research Site, Smiths Falls, Ontario
  - Research Site, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - Weekly CJC-1134-PC: CJC-1134-PC, 1.5 mg. weekly subcutaneous injection
- Arm 2 - Weekly CJC-1134-PC: CJC-1134-PC, start at 1.5 mg and titrate 0.5 mg weekly to 3-mg fixed weekly subcutaneous injection
- Arm 3 - Weekly CJC-1134-PC: CJC-1134-PC, start at 1.5 mg and titrate weekly to 2-, 2.5-, 3-, 3.5-, and 4.5-mg fixed weekly subcutaneous injection
- Arm 4 - Weekly CJC-1134-PC: CJC-1134-PC, start at 1.0 mg and titrate 1.0 mg weekly to 6.0-mg fixed weekly subcutaneous injection
- Arm 5 - Weekly Placebo: Weekly placebo for CJC-1134-PC administered weekly by subcutaneous injection
Period: Overall Study
Arm/Group | Arm 1 - Weekly CJC-1134-PC | Arm 2 - Weekly CJC-1134-PC | Arm 3 - Weekly CJC-1134-PC | Arm 4 - Weekly CJC-1134-PC | Arm 5 - Weekly Placebo
Started | 15 | 15 | 14 | 14 | 15
Completed | 12 | 14 | 11 | 13 | 14
Not Completed | 3 | 1 | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Weekly CJC-1134-PC | Arm 2 - Weekly CJC-1134-PC | Arm 3 - Weekly CJC-1134-PC | Arm 4 - Weekly CJC-1134-PC | Arm 5 - Weekly Placebo | Total
Number analyzed (Participants) | 15 | 15 | 14 | 14 | 15 | 73
Age, Customized [Count of Participants; unit: Participants]
  18 to 70 years | 15 | 15 | 14 | 14 | 15 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 6 | 8 | 4 | 31
  Male | 9 | 8 | 8 | 6 | 11 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Hemoglobin Change From Baseline (CFB) to Week 18
Time Frame: CFB to Week 18
Population: Completed Population
Measure: Mean (Standard Deviation); unit: Percent (%)
Arm/Group | Arm 1 - Weekly CJC-1134-PC | Arm 2 - Weekly CJC-1134-PC | Arm 3 - Weekly CJC-1134-PC | Arm 4 - Weekly CJC-1134-PC | Arm 5 - Weekly Placebo
Number analyzed (Participants) | 12 | 14 | 11 | 13 | 14
Percent (%) | -0.56 (0.597) | -0.56 (0.627) | -0.95 (0.746) | -0.95 (0.828) | -0.13 (0.811)

2. Secondary Outcome: Fasting Body Weight CFB to Week 18
Time Frame: CFB to Week 18
Population: Completed Population
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Arm 1 - Weekly CJC-1134-PC | Arm 2 - Weekly CJC-1134-PC | Arm 3 - Weekly CJC-1134-PC | Arm 4 - Weekly CJC-1134-PC | Arm 5 - Weekly Placebo
Number analyzed (Participants) | 12 | 14 | 11 | 13 | 14
kg | -1.91 (1.624) | -0.14 (4.122) | -1.37 (2.182) | -0.92 (1.999) | -1.85 (4.083)

3. Secondary Outcome: Time to Hyperglycemia Rescue
Time Frame: 18 weeks
Population: Completed Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1 - Weekly CJC-1134-PC | Arm 2 - Weekly CJC-1134-PC | Arm 3 - Weekly CJC-1134-PC | Arm 4 - Weekly CJC-1134-PC | Arm 5 - Weekly Placebo
Number analyzed (Participants) | 12 | 14 | 11 | 13 | 14
days | NA (NA) — 0 patient with hyperglycemia rescue | 47.0 (53.74) | NA (NA) — 0 patient with hyperglycemia rescue | NA (NA) — 0 patient with hyperglycemia rescue | 57.0 (NA) — Only 1 patient with hyperglycemia rescue

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | Arm 1 - Weekly CJC-1134-PC | Arm 2 - Weekly CJC-1134-PC | Arm 3 - Weekly CJC-1134-PC | Arm 4 - Weekly CJC-1134-PC | Arm 5 - Weekly Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15 | 0/13 | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15 | 0/13 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 3/12 | 11/15 | 8/13 | 8/13 | 5/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Weekly CJC-1134-PC (N=12) | Arm 2 - Weekly CJC-1134-PC (N=15) | Arm 3 - Weekly CJC-1134-PC (N=13) | Arm 4 - Weekly CJC-1134-PC (N=13) | Arm 5 - Weekly Placebo (N=14)
Nausea (Gastrointestinal disorders) | 1 | 7 | 5 | 6 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 1 | 1
Influenza like illness (General disorders) | 1 | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes